CLINICAL TRIAL: NCT04523181
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Proof of Concept Study to Evaluate the Safety and Efficacy of Antroquinonol in Hospitalized Patients With Mild to Moderate Pneumonia Due to COVID-19
Brief Title: Double-blind Study to Evaluate the Safety and Efficacy of Antroquinonol in Mild-Moderate COVID-19 Hospitalized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHCovid-2-001
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Covid-19
Keywords: Antroquinonol; COVID 19; pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — antroquinonol

STUDY DESIGN:
Intervention Model Description: A Phase 2 Randomized, Double blind, Placebo Controlled, Proof of Concept Study to Evaluate the Safety and Efficacy of Antroquinonol in Hospitalized Patients with Mild to Moderate Pneumonia due to COVID 19
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, Placebo Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Antroquinonol with SOC (Active Comparator): Antroquinonol in a dose of 100 mg (1 capsule) administered twice daily (BID) orally, for 14 days.
  Interventions: Drug: Antroquinonol
- Placebo with SOC (Placebo Comparator): Placebo (1 capsule) administered twice daily (BID) orally, for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antroquinonol — double-blind for antroquinonol and Placebo with same out-look and same frequency.
  Other Names: Hocena
  Arms: Antroquinonol with SOC
Other: Placebo — Capsule without active compound
  Arms: Placebo with SOC

SUMMARY:
To evaluate the safety and efficacy of antroquinonol treatment of mild to moderate pneumonia due to COVID-19, as measured by the proportion of patients alive and free of respiratory failure.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, Phase 2, proof of concept study in hospitalized patients with mild to moderate pneumonia due to COVID 19. Written informed consent must be obtained from all patients during screening. Following completion of all screening assessments and meeting of eligibility criteria, patients will either receive antroquinonol or placebo for 14 days in combination with SoC therapy per local SoC policies.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Male or female patients between 18 and 80 years of age.
3. Oxygen Saturation <94% in room air at screening.
4. Hospitalized with mild COVID 19 disease (not requiring oxygen therapy [WHO COVID-19 Clinical Improvement Ordinal Scale, score of 3] or requiring oxygen therapy by mask or nasal prong [WHO COVID-19 Clinical Improvement Ordinal Scale, score of 4]). Requirement of oxygen therapy by mask with reservoir to treat severe COVID 19 pneumonia is not allowed for enrollment.

   Note: Hospitalized patients can also include patients admitted to centers conditioned as hospitals to treat COVID-19 patients.
5. Chest x ray or computerized tomography (CT) scan consistent with pneumonia.
6. Onset of COVID-19 symptoms within 2 weeks prior to randomization.
7. Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV 2) infection confirmed by a polymerase chain reaction (PCR) test, antigen, or any authorized commercial or public health assay (nasopharyngeal, oropharyngeal, or respiratory samples, not serology testing).
8. Male patients and female patients of childbearing potential must agree to use protocol-specified methods of contraception.
9. Female patients of childbearing potential must have a negative pregnancy test at Screening or pretreatment on Day 1.
10. Male patients must agree not to donate sperm from the first dose through 90 days after the last dose of study treatment; female patients of childbearing potential should refrain from donation of ova from Day 1 until 90 days after the last dose of study treatment.
11. Patient is, in the opinion of the investigator, willing and able to comply with the study treatment regimen and all other study requirements.

Exclusion Criteria:

1. Female patient is pregnant or breastfeeding.
2. Any patient's concomitant life threatening condition, including but not limited to: requiring mechanical ventilation, acute respiratory distress syndrome, shock, or cardiac failure.
3. Evidence of multi lobar consolidation pneumonia or cavities on chest x ray or CT scan.
4. Severe COVID 19 disease as defined by the WHO COVID-19 Clinical Improvement Ordinal Scale, scores of 5 (non invasive ventilation or high flow oxygen), 6 (intubation and mechanical ventilation), or 7 (ventilation + additional organ support pressors, renal replacement therapy, ECMO).
5. Medical history significant for the following pulmonary diseases: lung cancer, cystic fibrosis, empyema.
6. Respiratory rate >30 respirations per minute.
7. History of abuse of drugs or alcohol that could interfere with adherence to study requirements, as judged by the investigator.
8. Treatment with other drugs thought to possibly have activity against COVID 19 within 7 days prior to enrollment or concurrently. Note: remdesivir or other authorized treatments for COVID 19 is allowed if considered SoC, if started prior to randomization or during the study.
9. Use of Antrodia camphorata -containing products within 2 weeks prior to the first administration of study drug.
10. Use of other investigational drugs within 30 days of dosing, or plans to enroll in another clinical trial of an investigational agent while participating in the present study. Note: authorized COVID 19 vaccines are not considered investigational and are not exclusionary.
11. Clinically significant abnormal electrocardiogram (ECG) at Screening, as determined by the investigator.
12. Patient requires frequent or prolonged use of systemic corticosteroids (≥20 mg of prednisone/day or equivalent for >4 weeks) or other immunosuppressive drugs (eg, for organ transplantation or autoimmune conditions).
13. Abnormal laboratory values at Screening:

    1. Estimated glomerular filtration rate <50 mL/min.
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 × upper limit of normal (ULN), or ALT/AST >3 × ULN plus total bilirubin >2 × ULN.
    3. Total bilirubin >1.5 × ULN, unless the patient has known Gilbert's syndrome.
    4. Hemoglobin <9 g/dL for females or <11 g/dL for males.
    5. Absolute neutrophil count <1,500/mm3.
    6. Thrombocytopenia (platelets count <100 × 109/L).
14. Treatment with any antiviral drugs (except remdesivir or other authorized treatments for COVID 19), or with any drugs known to be strong inducers or inhibitors of cytochrome P450 isoform (CYP) 2C19, CYP3A4, CYP2C8, and CYP2E1 within 14 days or 5 half lives prior to the start of study treatment. Drugs with a narrow therapeutic index that are substrates of 1A2, 2B6, 2C8, 2C9, 2C19, 3A, and 2D6 are also prohibited.
15. Inability to swallow oral medications or a gastrointestinal disorder with diarrhea (eg, Crohn's disease), malabsorption, or diarrhea of any etiology at baseline.
16. Any other clinically significant medical condition or laboratory abnormality that, in the opinion of the investigator, would jeopardize the safety of the patient or potentially impact patient compliance or the safety/efficacy observations in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (5):
  - Franciscan Health Michigan City, Michigan City, Indiana
  - Ascension.Via Christi Research, Wichita, Kansas
  - Adventist Healthcare Shady Grove Medical Center, Rockville, Maryland
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Duke University Southeastern Health, Lumberton, North Carolina
- Argentina (5):
  - Centro Gallego, Buenos Aires, Buenos Aires F.D.
  - Clinica de los Virreyes, Buenos Aires, Buenos Aires F.D.
  - Sanatorio Privado Mayo SA, Córdoba, Ciudad de Cordoba
  - Hospital Rawson, Córdoba, Cuidad de Cordoba
  - Clinica Viedma SA, Viedma, Pcia de Rio Negro
- Peru (5):
  - Clínica Internacional S.A. - Sede Lima, Lima Cercado, Lima region
  - Unidad de Investigacion, Hospital Nacional IV Alberto Sabogal Sologuren-Essalud, Red Assitencial Sabogal, Callao
  - Hospital de Chancay, Chancay
  - Asociación Civil Selva Amazónica, Iquitos
  - Hospital III Daniel Alcides Carrion - EsSalud, Tacna

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on October 15, 2020 and the last participant was enrolled on 08 OCT 2021.
Pre-assignment Details: Of 134 enrolled patients, 124 met inclusion criteria and 124 were randomized to treatment.
Period: Overall Study
Arm/Group | Antroquinonol With SOC | Placebo With SOC
Started | 62 (Patients Randomized) | 62 (Patients Randomized)
Treated (In the Antroquinonol with SOC group, 2 patients were randomized but not treated.) | 60 | 62
Completed | 54 (Completed Study) | 53 (Completed Study)
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Transferred to external facility. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antroquinonol With SOC | Placebo With SOC | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (11.75) | 50.2 (11.11) | 50.4 (11.39)
Age, Continuous [Median (Full Range); unit: years] | 50.5 [23 to 74] | 49.5 [24 to 75] | 50.0 [23 to 75]
Age, Customized [Count of Participants; unit: Participants]
  ≤65 years | 57 | 57 | 114
  >65 years | 5 | 5 | 10
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 35 | 30 | 65
  Female | 27 | 32 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 35 | 64
  Not Hispanic or Latino | 32 | 27 | 59
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 4 | 8
  White | 45 | 43 | 88
  More than one race | 6 | 13 | 19
  Unknown or Not Reported | 2 | 0 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.924 (8.0926) | 33.501 (7.2669) | 33.714 (7.6656)
BMI [Median (Full Range); unit: kg/m^2] | 30.487 [23.48 to 59.58] | 32.140 [22.99 to 59.52] | 31.250 [22.99 to 59.58]
Remdesivir or Other Authorized Treatments for COVID-19 Use [Count of Participants; unit: Participants] — Remdesivir or other authorized treatments for COVID-19 use at baseline.
  Participants
    Yes | 39 | 36 | 75
    No | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Recover Ratio
Description: Number of Patients Who are Alive and Free of Respiratory Failure (e.g., no need for invasive mechanical ventilation, non invasive ventilation, high flow oxygen, or ECMO) on Day 14.
Time Frame: 14 day
Population: The Intention-to-treat population (ITT). All randomized patients. Patients will be analyzed according to the treatment to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Antroquinonol With SOC | Placebo With SOC
Number analyzed (Participants) | 62 | 62
Participants
  Alive and Free of Respiratory Failure | 47 | 48
  Respiratory Failure | 1 | 0
  Missing | 14 | 14
  Death | 0 | 0

2. Secondary Outcome: Time to 2-point Improvement, Score 2 or Lower, and Score 0 From Baseline on the WHO COVID-19 Clinical Improvement Ordinal Scale
Description: Time to 2-point improvement from baseline, time to score 2 and lower from baseline and time to score 0 from baseline are measured by WHO COVID-19 Clinical Improvement Ordinal Scale
Time Frame: 28-day
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Antroquinonol With SOC | Placebo With SOC
Number analyzed (Participants) | 62 | 62
days
  Time to 2-point Improvement from Baseline | 7.0 [5.0 to 15.0] | 6.0 [5.0 to 9.0]
  Time to Score 2 or Lower from Baseline | 6 [4.0 to 10.0] | 6 [5.0 to 9.0]
  Time to Score 0 from Baseline | 29.0 [29.0 to 30.0] | 31 [30.0 to 42.0]

3. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization is the total number of days the patient is hospitalized during their participation in the study, up to Day 28.
Time Frame: 28 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo With SOC | Antroquinonol With SOC
Number analyzed (Participants) | 62 | 60
days
  Overall | 6.5 (5.54) | 6.4 (5.38)
  Age ≤65 Years Old: number analyzed (Participants) | 57 | 55
  Age ≤65 Years Old | 6.7 (5.72) | 6.4 (5.44)
  Age >65 Years Old: number analyzed (Participants) | 5 | 5
  Age >65 Years Old | 3.8 (1.10) | 6.8 (5.22)
  With COVID-19 Treatment at Baseline: number analyzed (Participants) | 36 | 39
  With COVID-19 Treatment at Baseline | 6.1 (5.71) | 5.1 (3.44)
  Without COVID-19 Treatment at Baseline: number analyzed (Participants) | 26 | 21
  Without COVID-19 Treatment at Baseline | 6.9 (5.38) | 9.0 (7.25)

4. Secondary Outcome: Time to Virological Clearance
Description: measured as study days from start of treatment to first negative SARS CoV 2 PCR test
Time Frame: 28 day
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Antroquinonol With SOC | Placebo With SOC
Number analyzed (Participants) | 62 | 62
days | 14.0 [6.0 to 15.0] | 15.0 [7.0 to 29.0]

5. Secondary Outcome: Number of Patients Who Recovered From Loss of Taste or Smell
Description: Patients with loss of taste or smell from baseline and back to normal during the observation period.
Time Frame: 28 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Antroquinonol With SOC | Placebo With SOC
Number analyzed (Participants) | 10 | 11
Participants | 10 | 8

ADVERSE EVENTS:
Time Frame: 4 Weeks
Description: In Antroquinonol with SOC group, 2 patients were randomized but not treated. All-Cause Mortality assessed for all randomized participants, Serious Adverse Events and Other (Not Including Serious) Adverse Events collected from randomized participants who got treated.
Arm/Group | Antroquinonol With SOC | Placebo With SOC
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 4/60 | 1/62
Other Adverse Events (participants affected / at risk) | 33/60 | 29/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antroquinonol With SOC (N=60) | Placebo With SOC (N=62)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antroquinonol With SOC (N=60) | Placebo With SOC (N=62)
Nausea (Gastrointestinal disorders) | 9 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Vomiting (Gastrointestinal disorders) | 8 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4
Blood lactate dehydrogenase increased (Investigations) | 2 | 1
Transaminases increased (Investigations) | 2 | 1
Blood bicarbonate decreased (Investigations) | 1 | 1
Blood cholesterol decreased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 1
Platelet count increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Rah (Skin and subcutaneous tissue disorders) | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Head discomfort (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Infusion site inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT04523181/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04523181/SAP_001.pdf